CLINICAL TRIAL: NCT00967564
Title: QUALITY OF LIFE ASSESSMENT IN PATIENTS AFFECTED BY MYELODYSPLASTIC SYNDROME
Brief Title: Survey on QUality of Life In myeloDisplasia (SQUID)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013075
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndrome; Quality of Life; Anemia; Epoetin alfa; Eprex
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Epidemiologic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: epidemiologic study QoL assessment
  Interventions: Other: epidemiologic study

INTERVENTIONS:
Other: epidemiologic study — QoL assessment

SUMMARY:
The purpose of this study is to evaluate the correlation between quality of life (QoL) and hemoglobin in patients affected by myelodysplastic syndrome and to compare the MDS (MyeloDisplastic Syndrome) patient's self-assessed QoL according to physician's evaluation

DETAILED DESCRIPTION:
In low-risk Myelodysplastic Syndrome (MDS), anemia is the major clinical problem and often represents the principal cause of symptoms which negatively influence quality of life (QoL). Moreover anemia has been associated with increased cardiac disease which, in older patients, may aggravate pre-existing conditions such as congestive heart failure. Patients with MDS often require red blood cell transfusions that further deteriorate patients' perception of well-being. This is an 18-month prospective observational investigation about the Quality of Life in Myelodysplastic patients with the aim to evaluate the correlation between hemoglobin (Hb) value and QoL and to compare the MDS patient's self-assessed QoL per physician's assessment. One hundred and fifty consecutive MDS patients at diagnosis and at least one with cytopenia - low level of hemoglobin or low level of neutrophils (a type of white blood cells that fights against infection) or low level of platelets (irregularly shaped cells found in blood that help prevent bleeding) - will be included in the evaluation. Demographic and disease-specific data will be collected and QoL will be evaluated by a specific questionnaire named QoL-E which will be completed both by patients and respective physicians. Study visits will be performed monthly until week 12; the subsequent visits will be performed at 6, 12 and 18 months. No Serious Adverse Event will be collected during the study, only adverse reaction to any Janssen-Cilag drug should be reported. This information may be important to optimize treatment according to patients' preferences and expectations, to detect functional complications, as well as to improve communication between patients and caregivers. Observational study - No study drug was administered.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary MDS
* At least one cytopenia according to International Prognostic Score System (IPSS) criteria (Hb < 10 g/dL
* Absolute neutrophils count (a type of white cell that fights against infection) < 1.800/µL
* platelets (irregularly shaped cells found in blood that help prevent bleeding) < 100.000/µL)
* Willing and able, based on investigator's judgment, to fill in QoL questionnaires

Exclusion Criteria:

* Refractory anemia with excess blasts (tumor cells located in the marrow > 20%)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) >3
* History of cerebrovascular disease with cognitive outcomes
* Psychiatric diseases or senile or vascular dementia
* Positive anamnesis for another clinically active tumor or when treatment has been stopped since less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Correlation between quality of life and hemoglobin in patients with new diagnosis of myelodysplastic syndrome | At baseline, at week 12, and at months 12 and 18

SECONDARY OUTCOMES:
Correlation between Hb changes and QoL changes | At baseline, at week 12, and at months 12 and 18 of observation
Comparison between the patient's and physician's QoL perception | At baseline, at week 12, and at months 12 and 18 of observation

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A. Clinical Trial, Study Director — Janssen-Cilag S.p.A.